CLINICAL TRIAL: NCT02270970
Title: Evaluation of Belimumab Impact on a BLyS Activity Signature Test in the Absence of Confounding Polypharmacy
Acronym: BLAST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMRF 14-18
Record Dates: First submitted 2014-10-13; First posted 2014-10-22 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Responders to Belimumab (Active Comparator): This Arm is defined as patients who complete 6 months of belimumab without and meet the primary endpoint
  Interventions: Biological: belimumab
- Non Responders to Belimumab (Active Comparator): This Arm is defined as patients who complete 6 months of study and do not meet the primary endpoint
  Interventions: Biological: belimumab

INTERVENTIONS:
Biological: belimumab — belimumab will be given at 10 mg/kg intravenously at Week 1, Week 2, Week 4 and monthly after that as was done in Phase III trials and approved in the FDA label
  Other Names: BenLysta

SUMMARY:
This will be an open label, non-randomized trial of belimumab in at least 20 subjects to test the feasibility of belimumab as a single agent and to capitalize on simplified background treatment regimens to determine immunologic differences between patients who do versus do not meet clinical response criteria.

DETAILED DESCRIPTION:
Primary Objective: This study will determine clinical response to belimumab using the SRI 4 (SLE Responder Index) which was used in the Phase III belimumab trials which led to its approval by the FDA. The population entered will be similar to the Phase III study population However, in this case background medications will be withdrawn at entry and brief steroid rescue with intramuscular depomedrol will provide immediate relief to cover the delay in belimumab effects. The co-primary objectives will be to determine time to disease flare compared to a historical control study (Biomarkers of Lupus Disease) and to determine whether more belimumab responders (defined by the SLE Responder Index) have a 50% decrease in the predefined BLAST signal (BlyS Activity Signal Test) than non-responders. This pilot study is not powered to draw firm conclusions about response rates in the absence of ongoing standard of care medications, but should 7-12 patients (of 20 completing the 6 month endpoint) meet the SRI response criteria, the feasibility of a larger, placebo controlled trial would be justified. The following instruments will be used to measure clinical lupus activity during the study: BICLA, SRI 5, changes in joint counts, global SLEDAI, BILAG, CLASI, PGA, and SF-36 and LFA-REAL measures.

The following are the definitions of these clinical outcome measures: SRI stands for SLE Responder Index which is a composite score comprised of a 4 (or alternatively 5) point decrease in the SLEDAI (SLE Disease Activity Index) coupled to no increase in the BILAG (British Isles Lupus Assessment Group) Index and no more than 10% increase in the Physician's Global Assessment. The global SLEDAI or BILAG is simply a comparison of the total SLEDAI or numerical composite BILAG score at baseline and after receiving belimumab. The CLASI refers to the Cutaneous Lupus Erythematosus Disease Area and Severity Index. the LFA REAL stands for the Lupus Foundation of America Rapid Evaluation of Activity in Lupus. The latter is a pilot instrument which will be tested in this study.

We will also integrate exploratory biologic discovery into the clinical trial to support both pre-specified and exploratory biomarker discovery. Data will be generated that might be used to help select more appropriate patient subsets for future trials and to guide optimal dosing strategies. Optimizing patient selection and dosing are important goals for further increasing demonstrable effect size in trials by increasing the response rates in the treatment groups. Thus, despite being a small pilot study, an ambitious goal is included to provide potential preliminary data conducive to optimize the use of belimumab. In general these analyses will also be descriptive, however our experience in the BOLD study suggests that comparing a group of 6-12 patients (presumed clinical response rate) who are enriched in expression of a particular biomarker vs a different group of 14-8 patients (defined in this case on basis of non-response to belimumab, or in the BOLD study by assignment to IFN high vs low subgroups) may, by virtue of representing different immunologic subsets of disease, produce statistically significant results in mean/median values of a number of biomarkers. More importantly, comparing "before and after" levels of BLyS and other cytokines may be quite sensitive to belimumab when it has clinical impact as well.

Obtaining this kind of preliminary data to better understand optimal patient selection could be a valuable approach to further increasing effect size in a future clinical trial. In fact, the two Parts of this project (single agent assessment and biomarker assessment) are co-dependent, since each increases the likelihood of interpretable data in patients with moderate severity. Indeed Part 2 would be less feasible without the strategy of Part 1 to decrease the conflicting immune signals of background medications, which have clouded interpretation of many treatments for SLE in the past.

Again, this will be an open label, six month study of belimumab treatment given to patients who qualify to receive this treatment under the United States labeling. Additionally, at entry to this study, patients must have a SLEDAI score of at least 6 which is identical to the disease activity minimum required for belimumab Phase III studies. Entry criteria will require results of a full clinical evaluation, CBC with differential, comprehensive metabolic profile (including liver function tests) and urinalysis (with reflex protein/creatinine ratio) prior to dosing.

The first dose will be given within 4 weeks of the screening visit and may take place as soon as the entry laboratories are returned. However, those patients who are stopping a major immune suppressant and/or those who require a steroid injection at entry will be encouraged to wait a minimum of 3 weeks before the initial belimumab dose. Blood samples for biomarkers (see below) will be drawn at the screening visit and just prior to the first dose to maximize disease assessment prior to steroid rescue as well as after withdrawal of background treatments. These will provide baseline data on the BLAST expression profile for each patient, which will be derived and standardized through the study of active SLE B Cells and in vitro B Cell gene expression responses to BLyS signaling. The highest BLAST signal recorded at either screening (prior to steroids) or baseline (after immune suppression withdrawal) will be employed as the baseline BLAST signal.

Subjects will be evaluated monthly by an investigator/subinvestigator who are trained for SLEDAI, BILAG 2004, and CLASI. Additional assays will be patient reported outcomes including the Short Form 36 (SF36) and the LFA REAL physician and patient endpoints. The co-primary clinical endpoint will be time to flare after the last steroid injection compared to the results of the BOLD study. The co-primary mechanistic endpoint will be measured at 3 months. This will be a comparison of rates of BLAST 50 response (50% decrease in fold change expression of BLAST panel genes as compared to healthy controls) in those who do or do not meet the clinical endpoint of SRI 4 without use of off-protocol medications. The SRI 4 endpoint will be met by meeting both the SRI criteria and no initiation of off- protocol immune suppressants or steroids. Although the stipulation of no off-protocol medications was not integrated into the initial definition of SRI it was required to meet the endpoint of the Phase III belimumab trials, since those who received off protocol treatments were removed from those studies and counted as non-responders. This brings our primary clinical endpoint in line with the intent of the primary endpoint in the Phase III belimumab studies. However our patients will not necessarily be removed from study for use of off protocol medications. After being designated a permanent non-responder in the primary endpoint such a patient might be further followed for exploratory analysis of improvement on additive medications.

This study will enroll patients until 20 have completed the protocol through the six month point. All patients will receive belimumab 10 mg/kg at baseline, 2 weeks later, 2 weeks after that and then q month. At each monthly visit history, physical, and blood tests (appropriate and as scheduled) to complete the outcome measures will be performed, and adverse event reporting and medication updates will be performed. Subjects may continue to take nonsteroidal anti-inflammatory medications (including prn NSAIDS) and up to 20 mg prednisone (or oral steroid equivalent) daily at screening and during the study although steroids will be tapered as tolerated. If the patient is taking hydroxychloroquine or an immune suppressant (e.g. mycophenolate mofetil, azathioprine, leflunomide, methotrexate, or a calcineurin inhibitor) at screening, these standard of care treatments must be stopped prior to the baseline visit, preferably a minimum of two weeks before baseline. Patients can elect to receive one or more depomedrol injection(s) up to a total of 320 mg total in individualized increments beginning at the time of the screening visit (if necessary) and/or up to and including the Month 2 visit. Daily oral steroids will be tapered as tolerated if and when the patient begins to improve.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet 1987 ACR criteria for SLE with 1996 modifications
2. SLEDAI >/= 6 at screening visit
3. Positive ANA OR anti-dsDNA within one year of screening
4. In the opinion of the investigator there is intent to treat with a biologic (e.g. patient failed standard of care treatment) however there is no organ threatening disease

Exclusion Criteria:

1. Hg less than 8.0 or hemolytic anemia
2. Lymphocyte count less than 0.4
3. AST/ALT greater than 2.5 times ULN
4. Infection requiring IV antibiotics within a month of screening or oral antibiotics within two weeks of first dose
5. Active chronic infections (such as tuberculosis) which have not been treated or tb exposure in a person under 40 who has not received suppressive therapy for at least 3 months. Herpes zoster outbreak within three months of dosing. (Suppressive therapy for herpes simplex is not an exclusion criterion).
6. Cancer within 5 years (except for completely excised cervical carcinoma in situ or excised non-melanoma skin cancer)
7. Inability or unwillingness to follow the protocol
8. If WOCBP, inability or unwillingness to practice an acceptable method of contraception (including abstinence, barrier method with spermicide, or hormonal treatment
9. Inability or unwillingness to withdraw from hydroxychloroquine and/or any immune suppressive therapy being taken despite option for immediate steroid treatment and later treatment rescues as needed.
10. Any illness or condition that, in the opinion of the investigator, would cause undue hardship or risk to the subject by participating in the protocol

    -

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
BLAST-50 response rate in clinical responders vs non responders | 3 months
  The BLyS Activity Signature Test will determine the rate at which pre-specified biomarkers of BLyS signaling in B Cells are reduced at least 50% in those who do or do not meet the SRI-4 clinical response criteria (the latter defined as a decrease in the SLE Disease Activity Index (SLEDAI) of 4 or more points, no increase in the BILAG index of disease activity, no more than a 10% increase in Physician's Global Assessment and no rescue medications after Month 2

SECONDARY OUTCOMES:
Time to flare compared to historical (untreated) controls from the BOLD study | 6 months
  The patients taking part in the BOLD study were in a very similar protocol but without an interventional study medication once the steroids were given. 75% flared within 4 months and 97.6% flared within 6 months of the last steroid shot. Thus they can serve as historical controls of some value in this study which does not include a placebo group. Flare will be defined, as in the BOLD study as an increase in SLEDAI of 4 or more points or one grade worsening in at least one BILAG-defined score, also requiring the clinician's determination of a clinically significant worsening and intention to treat
SRI-4 response rates compared to historical controls from the BOLD study | 6 months
  The SRI-4 is identical to the SRI-4 described in the primary endpoint
SRI-5 response rates compared to historical controls from the BOLD study | 6 months
  The SRI-5 is identical to the SRI-4 described in the primary endpoint except that it requires at least a 5 point improvement in the SLEDAI. The BICLA (BILAG-based Combined Lupus Assessment) requires one grade of improvement in every BILAG score present at baseline along with no worsening in any BILAG or SLEDAI descriptor, no more than a 10% worsening by Physician's Global Assessment and no further rescue treatment after 2 months
BICLA response rates compared to historical controls from the BOLD study | 6 months
  The BICLA (BILAG-based Combined Lupus Assessment) requires one grade of improvement in every BILAG score present at baseline along with no worsening in any BILAG or SLEDAI descriptor, no more than a 10% worsening by Physician's Global Assessment and no further rescue treatment after 2 months
Tender and swollen joint counts at baseline and each month | 6 months
  Joint counts will be performed using the ACR 28 joint count format
PGA at baseline and each month | 6 months
  PGA stands for Physician's Global Assessment which is a 100mm scale based on the SELENA SLEDAI version of the PGA which includes landmarks for mild, moderate and severe disease activity
CLASI at baseline and each month | 6 months
  This is a scoring system for mucocutaneous manifestations of lupus segmented by area of the body and severity
LFA-REAL at baseline and each month | 6 months
  This is a series of scales based on the SELENA SLEDAI PGA which breaks down the assessment by organ system and includes assessments by both clinicians and patients

OTHER OUTCOMES:
Exploratory Biomarker Studies | 6 months
  To be determined because it will be exploratory
Descriptive Safety Data | 6 months
  Serious Adverse Events, all Adverse Events and Adverse Events of Special Interest will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Thanou, M.D., Principal Investigator — Oklahoma Medical Research Foundation
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided